CLINICAL TRIAL: NCT03827278
Title: Human Immunodeficiency Virus Negative Host Talaromyces Between Voriconazole and Amphotericin B Sequential Itraconazole Therapy
Brief Title: Comparative Study of Human Immunodeficiency Virus Negative Host Talaromyces Between Voriconazole and Amphotericin Sequential Itraconazole Therapy
Acronym: CSHHTVASIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The Fourth People's Hospital of Nanning (Other); Guilin Medical College (Other); Nanning Second People's Hospital (Other)
Responsible Party: Principal Investigator, Qiu Ye, Clinical Professor, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSM-AMB-VOR-2018
Record Dates: First submitted 2019-01-25; First posted 2019-02-01 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Talaromyces in Human Immunodeficiency Virus Negative; To Compare Voriconazole and Amphotericin Sequential Itraconazole Therapy; To Dynamically Monitor the Anti-Interferon-γ Autoantibodies
Keywords: Talaromyces; voriconazole; Amphotericin Sequential Itraconazole therapy; anti-Interferon-γ autoantibodies
MeSH Terms: interventions — Voriconazole; Amphotericin B; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV Negative Host talaromyces using Voriconazole (Experimental): Voriconazole On the first day, 6 mg/kg bid was given, and then 4 mg/kg bid was given intravenously for 6 days, and then oral voriconazole 200 mg bid was administered to maintain treatment for at least 6 months.
  Interventions: Drug: Voriconazole
- HIV Negative talaromyces AMB Sequential Itraconazole (Experimental): Amphotericin B (AMB) sequential itraconazole group (intravenous amphotericin, dose 0.7 - 1.0 mg / kg / d, 14 days, then changed oral itraconazole 200 mg bid for 10 weeks, after which 100 mg bid maintenance Until cluster of differentiation 4 (CD4+ T) cells are greater than 100 cells/L for at least 6 months
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — 6mg/kg bid, was given on the first day, followed by intravenous 4mg/kg bid for 6 days, followed by oral Valconazole 200mg bid for at least 6 months.
  Amphotericin B sequential itraconazole group (intravenous amphotericin, dose 0.7 - 1.0 mg / kg / d, 14 days, then changed oral itraconazole 200 mg bid for 10 weeks, after which 100 mg bid maintenance Until CD4+ T cells are greater than 100 cells/L for at least 6 months
  Other Names: Amphotericin; Itraconazole

SUMMARY:
Through a multi-center large-sample non-randomized controlled study, the effect of voriconazole, amphotericin B sequential itraconazole therapy on Talaromyces in Human Immunodeficiency Virus（HIV）negative hosts were compared to clarify whether the two therapies were equivalent; A comprehensive efficacy evaluation system and standard treatment program was established to provide a basis for standardized treatment of Talaromyces in Human Immunodeficiency Virus negative hosts.The observational indicators included: 2-week all-cause mortality; 24-week all-cause mortality; clinical improvement time; level of decrease of fungus in the blood culture medium two weeks before treatment; recurrence; appearance of adverse drug reaction at the level 3 and above. Dynamically monitor the immune cells and factors like anti-Interferon-γ autoantibodies, Interferon-γ, Th1/Th2, and Th17/Treg in the HIV-negative Talaromyces host microenvironment, and observe the host's immune status and its change. 3. study the effect of absence of Interferon-γ and Interferon-γ Receptor (IFN-γR）on the activation and function of anti-Interferon-γ autoantibodies, Th1/Th2, and Th17/Treg by establishing a Talaromyces mouse model that knocks out the Interferon-γ and IFN-γR gene and a IFN-γ silenced cell model; Study the effect of anti-IFN-γ autoantibody on the activation and function of IFN-γ、Th1/Th2、Th17/Treg by increasing its titer in vitro and vivo; determine by which path the anti-IFN-γ autoantibody of HIV-negative host influences its immune regulation mechanism; finally, the intervention effect of IFN-γ on high titer anti-IFN-γ autoantibodies is studied, providing a new idea for immunotargeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-negative adults (≥18 years of age) who diagnosis of talaromyces that was confirmed by either microscopy or culture
2. Must be able to swallow tablets

Exclusion Criteria:

1. Pregnancy, central nervous system involvement assessed either clinically or by analyses of cerebrospinal fluid
2. An allergy to voriconazole, itraconazole or amphotericin
3. The concomitant use of certain medications that interact with voriconazole, itraconazole or amphotericin
4. An alanine aminotransferase or aspartate aminotransferase level of more than 400 U per liter
5. An absolute neutrophil count of less than 500 per cubic millimeter
6. A creatinine clearance of less than 30 ml per minute (calculated by the method of Cockcroft and Gault)
7. a concurrent diagnosis of cryptococcal meningitis
8. concurrent treatment with rifampicin
9. previous treatment for talaromyces for more than 48 hours
10. HIV positive who diagnosis of talaromyces.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-30 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with all-cause mortality | up to 2 weeks
  defined as the absolute risk of death from any cause during the first 2 weeks
Number of Participants with all-cause mortality | up to 24 weeks
  defined as the absolute risk of death from any cause during 24 weeks
Number of Participants with Clinical resolution of talaromyces | 3 days
  Clinical resolution of talaromyces was defined as a temperature of less than 38°C (100°F) for 3 days, resolution of skin lesions, and tertile blood cultures. Early fungicidal activity was defined as the rate of decline in blood T. marneffei colony forming units (CFUs).
Number of Participants with Early fungicidal activity | up to 2 weeks
  defined as the rate of decline in blood T. marneffei CFUs from sterical blood cultures obtained during the first 2 weeks.
Number of Participants with Relapse of talaromyces | an average of 1 year
  defined as the recurrence of symptoms and a positive fungal culture from any sterile site that led to reinduction of therapy in patients who had achieved clinical resolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Le T, Kinh NV, Cuc NTK, Tung NLN, Lam NT, Thuy PTT, Cuong DD, Phuc PTH, Vinh VH, Hanh DTH, Tam VV, Thanh NT, Thuy TP, Hang NT, Long HB, Nhan HT, Wertheim HFL, Merson L, Shikuma C, Day JN, Chau NVV, Farrar J, Thwaites G, Wolbers M; IVAP Investigators. A Trial of Itraconazole or Amphotericin B for HIV-Associated Talaromycosis. N Engl J Med. 2017 Jun 15;376(24):2329-2340. doi: 10.1056/NEJMoa1613306. PMID 28614691
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28614691